CLINICAL TRIAL: NCT06888167
Title: Experimental, Drug-free, Cross-sectional, Single-centre Study to Assess the Association Between Metabotypes of Dietary (poly)phenols and Beta-cell Mass and Function.
Brief Title: Food (poly)phenol Metabotypes and Beta-cell Mass and Function.
Acronym: META-BETA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: University of Parma (Other)
Responsible Party: Principal Investigator, Alessandra Dei Cas, Prof., Azienda Ospedaliero-Universitaria di Parma
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 683-2023
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Participants in the OPCT study - MT 'A', low disposition index (n=10) (Other)
  Interventions: Other: Study setting
- Participants in the OPCT study - MT 'A', high disposition index (n=10) (Other)
  Interventions: Other: Study setting
- Participants of the OPCT study - MT 'B', low disposition index (n=10) (Other)
  Interventions: Other: Study setting
- Participants of the OPCT study - MT 'B', high disposition index (n=10) (Other)
  Interventions: Other: Study setting

INTERVENTIONS:
Other: Study setting — The subjects in the study will undergo two days of visits, in random order.
  1. Following a fasting period of at least 4 hours, the study participants will undergo a PET-CT examination with Ga-exadin-4. Fasting will reduce the endogenous secretion of GLP-1 by the small intestine, which can otherwise compete with exendin-4 for binding to GLP-1R. Blood glucose will be measured before the injection of the tracer and monitored at each time point.
  2. On a fasting basis, the anthropometric data of the enrolled subjects will be collected and they will undergo a short interview on their lifestyle. Subsequently, at time 0, the subjects will ingest a standard mixed meal consisting of 2 commercially available "ABC Parmareggio" snacks. Venous blood samples will be taken at specific time intervals (from -20 to 300 minutes) to measure glucose, C-peptide, insulin, glucagon, GLP-1 and glucose-dependent insulinotropic (GIP) curves. An additional blood sample will be taken at time -10 in order to isolate

SUMMARY:
Cross-sectional, single-centre, 'low intervention' clinical study, without drug or medical device testing, with low-risk diagnostic technique.

DETAILED DESCRIPTION:
Chronic diseases, such as cardiovascular diseases (CVD) and cardiometabolic diseases (CMD), including type 2 diabetes (DT2), represent one of the most important public health problems. Lifestyle intervention can help prevent or delay the development of diabetes mellitus. In this regard, several nutritional guidelines have been developed to promote cardiovascular and metabolic health. These recommendations promote regular consumption of fruit and vegetables, whole grains, healthy sources of protein; foods that are particularly rich in polyphenols, with known health benefits. However, their application to improve cardiometabolic health is hampered by the heterogeneity of individual response to the consumption of dietary (poly)phenols. In an intervention study entitled 'Aggregate Metabolic Phenotypes for (Poly)Phenols: Development of an Oral (Poly)Phenol Challenge Test (OPCT)', the variability of the urinary concentration of phenolic metabolites among 300 volunteers after consumption of (poly)phenol-rich tablets was assessed and predictive algorithms were generated to identify and group individuals with similar metabolic/phenotypic profiles (metabotyping). The role of these specific metabotypes (MTs) on cardiometabolic health and, more specifically, on human pancreatic beta-cell function (BCF) and mass (BCM) of individuals remains to be explored. Identifying, in fact, an association between different MTs and a higher/lower BCM/BCF would allow to evaluate the potential risk of individuals to develop metabolic diseases, as well as to act with dietary interventions aimed at protecting and preventing possible damage to pancreatic beta-cells.

In this study "Food (poly)phenol Metabotypes and Beta-cell mass ad function" (META-BETA), we intend to address - specifically - the effects on a tissue fundamental for metabolic health, namely pancreatic beta-cells. To achieve this goal, the investigators intend to focus on the action of active molecules derived from food (poly)phenols, on the function and mass of pancreatic beta-cells. In order to take into account interindividual differences, they will also explore the effects of specific metabolites derived from (poly)phenols in beta-cells derived from individuals with opposite MTs and Disposition Index, previously identified in the OPCT study.

The project is divided into two parts:

1. Association study: the association between different MTs and disposition index was explored in 300 healthy adult subjects, previously enrolled in the OPCT study. In four paired subgroups (n=10), recruited in two opposite MTs and with maximum difference in disposition index, BCFxM will be evaluated with a mixed meal complete with all macronutrients in a balanced way. In addition, BCM will be measured with the PET-CT method (beta-cell specific radioligand, Ga-exendin-4). The ratio between BCFxM (MMTT) and BCM (PET-CT) will provide the in vivo BCF data. Furthermore, during a short interview, data on the lifestyle of the subjects in the study will be collected.
2. Cause-effect study: Induced pluripotent stem cells (iPSCs), derived from peripheral blood mononuclear cell (PBMCs), from 2 subjects matched for each MT, with different BCF and BCM, will be differentiated into beta-cells where the effects of polyphenol metabolites will be evaluated. Experiments will be conducted both in control conditions and in the presence of lipotoxicity induced by stearic acid (SA).

The primary objective of this study is therefore to identify specific metabotypes (MTs) that are associated with different pancreatic beta-cell mass and function (BCFxM).

ELIGIBILITY:
Inclusion Criteria:

* Having been enrolled in the OPCT study;
* Ability to understand the methods, purposes and implications of the study, and to give free and informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Previous exposure to ionizing radiation in research programs;
* History of psychiatric illness or alcohol abuse;
* Head trauma;
* Active neurological disease;
* Claustrophobia;
* Active malignant neoplastic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Specific metabotypes (MTs) that associate with different pancreatic beta-cell mass and function (BCFxM). | through study completion, an average of 3 months after enrolment
  BCFxM=parametes derived from mixed meal test Beta cell function (BCF)=BCFxM/BCM

SECONDARY OUTCOMES:
Pancreatic beta cell mass (BCM) | through study completion, an average of 3 months after enrolment
  Beta cell mass index (BCM)=68GA-exendin-4-Standard Uptake Value (SUV)*pancreatic volume
Pancreatic beta cell function (BCF) | through study completion, an average of 3 months after enrolment
  BCFxM/BCM
Specific MTs that exhibit different beta-cell mass (BCM) in vivo. | through study completion, an average of 3 months after enrolment
Personalized nutritional interventions. | through study completion, an average of 3 months after enrolment
  Lay the foundation for the design of personalized nutritional interventions that can reduce the risk of specific diseases, such as the risk of developing type 2 diabetes and the consequences of diabetes-related organ damage (including cardiovascular system) depending on one's MT.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria di Parma, Parma, PR, Italy

REFERENCES:
- [Background] Rezania A, Bruin JE, Arora P, Rubin A, Batushansky I, Asadi A, O'Dwyer S, Quiskamp N, Mojibian M, Albrecht T, Yang YH, Johnson JD, Kieffer TJ. Reversal of diabetes with insulin-producing cells derived in vitro from human pluripotent stem cells. Nat Biotechnol. 2014 Nov;32(11):1121-33. doi: 10.1038/nbt.3033. Epub 2014 Sep 11. PMID 25211370
- [Background] Blanchi B, Taurand M, Colace C, Thomaidou S, Audeoud C, Fantuzzi F, Sawatani T, Gheibi S, Sabadell-Basallote J, Boot FWJ, Chantier T, Piet A, Cavanihac C, Pilette M, Balguerie A, Olleik H, Carlotti F, Ejarque M, Fex M, Mulder H, Cnop M, Eizirik DL, Jouannot O, Gaffuri AL, Czernichow P, Zaldumbide A, Scharfmann R, Ravassard P. EndoC-betaH5 cells are storable and ready-to-use human pancreatic beta cells with physiological insulin secretion. Mol Metab. 2023 Oct;76:101772. doi: 10.1016/j.molmet.2023.101772. Epub 2023 Jul 11. PMID 37442376
- [Background] Eriksson O, Velikyan I, Haack T, Bossart M, Laitinen I, Larsen PJ, Berglund JE, Antoni G, Johansson L, Pierrou S, Tillner J, Wagner M. Glucagonlike Peptide-1 Receptor Imaging in Individuals with Type 2 Diabetes. J Nucl Med. 2022 May;63(5):794-800. doi: 10.2967/jnumed.121.262506. Epub 2021 Sep 9. PMID 34503957